CLINICAL TRIAL: NCT03415113
Title: Impact of Medication Reconciliation at Discharge on Potentially Inappropriate Medications in the Elderly : Community-hospital Coordination. ICM2SA
Brief Title: Impact of Medication Reconciliation at Discharge on Potentially Inappropriate Medications in the Elderly : Community-hospital Coordination
Acronym: ICM2SA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2016_843_0003
Record Dates: First submitted 2017-12-27; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Hospital; Geriatric
Keywords: Medication reconciliation at discharge, potentially inappropriate medications, elderly.

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The geriatric population is exposed to poly-medication. Furthermore, old people have important pharmacodynamic and pharmacokinetic changes that expose to much drug iatrogenic. Adverse drug effects are a great cause for hospitalization that is why the knowledge of the complete list of medications taken by the patient is necessary. The poly-medication in elderly can lead to extremely serious clinical consequences and significant costs. Reference documents specific to geriatrics guide the doctor in therapeutic choices. On the one hand, the Laroche's criteria lists all PIM of the French pharmacopoeia in elderly. On the other hand, STOPP/START criteria are a tool for detect PIM listing inappropriate drugs and criteria of potentially drug omissions. This has been validated in French language. It is important that any changes proposed by the geriatrician resulting in just prescription is sustainable beyond the hospitalization to prevent the recurrence of adverse effects. Effective community-hospital coordination is essential.

Medication reconciliation is defined as the formal process of checking the complete, accurate list of a patient's previous medication - including drug name, dosage, frequency, and route - and comparing it with the prescription after a transition of care (on admission, after transfer to another medical unit, and/or at discharge).

Two groups of patients will be created, one for which medication reconciliation at discharge will be practiced and the other a similar process but not standardized. Four to eight weeks after the discharge, the member of the pharmacy team is calling the usual community pharmacy to get the first non-hospital prescription by fax and compare the number of PIM with the prescription before hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 75 years
* Pharmaceutical interview at the medication reconciliation at admission in Geriatrics Acute Care Unit.
* ≥ one PIM on the prescription before admission
* Identification of the usual referent community pharmacist
* Output of the unit by a return home
* Affiliation to a social security scheme

Exclusion Criteria:

* Patients undergoing a regime of legal protection.
* Patients unable to cooperate in pharmaceutical interview at the medication reconciliation at admission whatever reason.
* Refusal to participate in the study.
* Output of the unit by transfering to another care unit or death

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Geriatic population
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Quantification of potentially inappropriate medication prescription | 4 or 8 weeks
  Quantification of potentially inappropriate medication on the first non-hospital

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume DESCHASSE, MD, Principal Investigator — CHU Amiens